CLINICAL TRIAL: NCT03279549
Title: A Randomized, Controlled, Prospective Clinical Trial on the Key Technology of Burn Wound Treatment
Brief Title: Research on the Key Technology of Burn Wound Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); Ruijin Hospital (Other); Southwest Hospital, China (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Hu Dahai, Director of Burn Center, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20140709-1
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Fibroblast Growth Factor 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- dressing change group (Active Comparator): Routine dressing change group
  Interventions: Procedure: Routine dressing change
- Dermal matrix dressing group (Experimental): Limited debridement & Acellular dermal matrix dressing group.
  Interventions: Procedure: Limited debridement & Acellular dermal matrix dressing
- Epidermal cell spraying group (Experimental): Limited debridement & Epidermal cell spraying group
  Interventions: Procedure: Limited debridement & Epidermal cell spraying
- BFGF group (Experimental): Limited debridement & Basic fibroblast growth factor group
  Interventions: Procedure: Limited debridement & Basic fibroblast growth factor

INTERVENTIONS:
Procedure: Routine dressing change — Through regular dressing changes to clean the wound, reduce bacterial growth in the wound and protect the wound. In recent years, nano-silver ion gel and dressings are widely used in burns, which effectively reduced the risk of wound infection and beneficial for wound healing. This technique is widely used in clinic.
  Arms: dressing change group
Procedure: Limited debridement & Acellular dermal matrix dressing — In the removal of necrotic dermis in the "rather not deep" principle, as far as possible not damage the normal dermal tissue and skin accessories. This could improve circulation of wounds and improve wound healing. The xenogeneic acellular dermal matrix dressing has a better protective effect on burn wound after debridement. After covering, the wound will remain alive for about two weeks, providing a good microenvironment for wound repair.
  Arms: Dermal matrix dressing group
Procedure: Limited debridement & Epidermal cell spraying — In the removal of necrotic dermis in the "rather not deep" principle, as far as possible not damage the normal dermal tissue and skin accessories. This could improve circulation of wounds and improve wound healing. Epidermal cell spraying technology is a brand new method to rapidly collect epidermal cells from patients themselves and then used on their wounds. The recipient site is 40-80 times than the donor site.
  Arms: Epidermal cell spraying group
Procedure: Limited debridement & Basic fibroblast growth factor — In the removal of necrotic dermis in the "rather not deep" principle, as far as possible not damage the normal dermal tissue and skin accessories. This could improve circulation of wounds and improve wound healing. BFGF is a kind of polypeptide capable of promoting the growth of fibroblasts, and it also promotes the proliferation, differentiation and migration of epidermal cells. Studies have shown that bFGF could significantly improve the healing of burn wounds.
  Arms: BFGF group

SUMMARY:
Burns are common injuries in the daily life and wars. With the development of medical techniques, the mortality has been significantly reduced. However, the deformity and disability caused by hypertrophic scar have not been improved effectively since the wound repair technology is limited and controversial, especially on the early treatment of deep second degree burns. The prognosis of burns is of great difference. In recent years, the promotion of wound repairing technologies provides a new opportunity for improving the quality of wound healing and solving the problem of scar formation. Although some new methods and techniques have shown significant efficacy in clinic, clinical researches with large samples conducted in multiple centers are still deficient, impeding the evaluation of their superiority. Therefore, the current protocol focuses on the repair of deep second degree burns based on previous researches. There are four types of treatment protocols for wounds. Patients were divided into four groups randomly, including regular dressing change group, controlled debridement + biological dressing covering group (xenogeneic acellular dermal matrix), controlled debridement + epidermal cell cultivation group, controlled debridement + bFGF treatment group. The wound healing rate, healing time and scar formation were observed. The availability and security were evaluated. Further more, treatment guidelines and expert consensuses on deep second degree burn wounds were concluded. Above studies are important to promote the treatment of deep second degree burns to be scientific, standardized and professional in China.

ELIGIBILITY:
Inclusion Criteria:

1. Area of deep second burn wound >=10cm×10cm，total burn area ≤50% TBSA.
2. Within 96 hours after burns and could be managed within 24 hours after included.
3. Ages from 18 to 60.
4. No serious breathing, circulation and other systemic diseases, no surgical contraindications.
5. Agrees to participate in this trial and has signed an informed consent form.

Exclusion Criteria:

1. Have severe inhalation injury or shock, or acute respiratory failure；
2. There are serious heart (especially the recent myocardial infarction, myocardial damage, etc.), brain, liver, kidney, lung and other organ disease;
3. Susceptible to allergies；
4. Islamic believers
5. Pregnant women
6. Other cases that are not suitable for study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | 21 days after treatment
  Healing time is the number of days when the wound healed completely after management.

SECONDARY OUTCOMES:
Wound healing rate | 21 days after treatment
  Wound healing rate =（area before management - area after management）/ area before management×100%.
Scar formation | 6 months after treatment
  Vancouver scar score

CONTACTS AND LOCATIONS:
Overall Officials: Xie Songtao, Doctor, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: No